CLINICAL TRIAL: NCT05639218
Title: Impact of Optimal Pharmacotherapy on Plasma Lipid Profile and Qualitative Features of Atherosclerotic Plaques in Very-high Cardiovascular Risk Patients With Established Atherosclerotic Cardiovascular Disease
Brief Title: Impact of Optimal Pharmacotherapy on Lipid Profile and Qualitative Features of Atherosclerotic Plaques
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pauls Stradins Clinical University Hospital (Other)
Responsible Party: Principal Investigator, Karlis Trusinskis, MD, Pauls Stradins Clinical University Hospital
Other Study IDs: PCSK9I-0621
Record Dates: First submitted 2022-11-23; First posted 2022-12-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Atherosclerotic Cardiovascular Disease
Keywords: Atherosclerosis; PCSK9; Inclisiran; NIRS-IVUS; LDL-C
MeSH Terms: conditions — Atherosclerosis | interventions — ALN-PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Inclisiran — Patients are receiving PCSK9 inhibitors or inclisiran in the context of optimal hypolipidemic pharmacotherapy
  Other Names: PCSK9 inhibitor

SUMMARY:
Lipid accumulation, with mostly emphasized role of low-density lipoprotein cholesterol (LDL-C), is the pathogenetic cornerstone of atherosclerotic cardiovascular disease. Standard hypolipidemic therapy, based on statins and ezetimibe, does not always decrease LDL-C levels enough to achieve therapeutic goals. A novel and promising direction is inhibition of proprotein convertase subtilisin/kexin type 9 (PCSK9) in hepatocytes, subsequently reducing LDL-C receptor degradation and increasing intracellular LDL-C uptake.

Aim of this study is to evaluate the effect of optimal hypolipidemic pharmacotherapy, including PCSK9 inhibitors and inclisiran, on plasma lipid profile and qualitative features of atherosclerotic plaques in very-high cardiovascular risk patients.

This study enrolls patients with an established atherosclerotic cardiovascular disease, receiving PCSK9 inhibitors or inclisiran as add-on treatment to statins in maximally tolerated dose and/or ezetimibe.

Effect of hypolipidemic pharmacotherapy is evaluated by analysis of plasma lipid profile parameter changes and qualitative features of atherosclerotic plaques using Near-Infrared Spectroscopy Intravascular Ultrasound Imaging (NIRS-IVUS) method.

Results of the study would be sufficient for complementing evidence regarding therapeutic strategy in very-high cardiovascular risk patients.

DETAILED DESCRIPTION:
Background:

Lipid accumulation in artery walls is the pathogenetic cornerstone of atherosclerosis. The most commonly studied risk factor of atherosclerotic cardiovascular disease is low-density lipoprotein cholesterol (LDL-C), nevertheless other plasma lipids have an established role as well. LDL-C is considered the primary target for cardiovascular risk reduction, with therapeutic goal <1.4 mmol/l in very-high cardiovascular risk patients with established atherosclerotic cardiovascular disease. Standard hypolipidemic therapy, based on statins and ezetimibe, is not always effective enough. Novel and promising direction is proprotein convertase subtilisin/kexin type 9 (PCSK9) - protease that binds LDL receptors in hepatocytes, subsequently promoting their lysosomal degradation. This process leads to reduced intracellular LDL-C uptake and increased LDL-C concentration in plasma. PCSK9 inhibitors - monoclonal antibodies evolocumab and alirocumab are successfully used in clinical practice, with a proven effectiveness in clinical trials ODYSSEY and FOURIER. An innovative medication is inclisiran - small interfering ribonucleic acid (siRNA) molecule that interferes with translation of messenger RNA (mRNA) of PCSK9 in hepatocytes as a result of complementary binding. Subsequently levels of synthesized PCSK9 are reduced, resulting in positive impact on plasma lipid profile. Inclisiran has demonstrated remarkable efficacy and safety profile in ORION clinical trials, being registered in European Medicines Agency since year 2020. Real-world data regarding optimal lipid-lowering pharmacotherapy, including experience with new medications, is of great clinical interest, studying effect on plasma lipid profile, as well as qualitative features of atherosclerotic plaques using Near-Infrared Spectroscopy Intravascular Ultrasound Imaging (NIRS-IVUS) method.

Aim:

Aim of this study is to evaluate effect of optimal hypolipidemic pharmacotherapy on plasma lipid profile and and qualitative features of atherosclerotic plaques in very-high cardiovascular risk patients receiving PCSK9 inhibitors or inclisiran as add-on treatment to statins in maximally tolerated dose and/or ezetimibe.

Study design:

Prospective observational study.

Study population:

Very-high cardiovascular risk patients with an established atherosclerotic cardiovascular disease, receiving PCSK9 inhibitors or inclisiran as add-on treatment to statins in maximally tolerated dose and/or ezetimibe in the context of optimal hypolipidemic pharmacotherapy, in whom NIRS-IVUS investigation has been performed.

Data acquisition:

Patients fulfilling eligibility criteria and agreeing to participate in the study are included. Baseline demographic and medical data is acquired, with subsequent follow-up ambulatory visits after 3 and 6 months after PCSK9 inhibitor or inclisiran therapy initiation. After 15 months since inclusion, follow-up with NIRS-IVUS performed is foreseen. For analysis of obtained data MS Excel and IBM SPSS Statistics software is used.

Clinical implications:

Results of this study would be of high clinical interest for complementing evidence and improving outcomes regarding therapeutic strategy in very-high cardiovascular risk patients with an established atherosclerotic cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Very high cardiovascular risk - documented atherosclerotic cardiovascular disease
* On maximally tolerated statin and/or ezetimibe therapy for at least 1 month LDL-C treatment target <1.4 mmol/l not achieved
* Receiving PCSK9 inhibitor or inclisiran as add-on treatment to maximally tolerated statin dose and/or ezetimibe in the context of optimal pharmacotherapy
* NIRS-IVUS performed (written informed consent for the procedure signed according to regulations in the hospital)
* Available blood test results - plasma lipid profile
* Patient agrees to participate in the study (signed informed consent)

Exclusion Criteria:

* Not fulfilling any of inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study enrolled very high cardiovascular risk patients with established atherosclerotic cardiovascular disease, who receive PCSK9 inhibitors or inclisiran as add-on treatment to maximally tolerated statin dose and/or ezetimibe in the context of optimal pharmacotherapy, and in whom NIRS-IVUS has been performed in the Latvian Centre of Cardiology, Pauls Stradins Clinical University Hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
LDL-C level | 15 months
  Plasma LDL-C level changes in patients receiving PCSK9 inhibitors or inclisiran
Qualitative features of atherosclerotic plaques | 15 months
  Changes in qualitative features of atherosclerotic plaques assessed by NIRS-IVUS investigation

CONTACTS AND LOCATIONS:
Overall Officials: Karlis Trusinskis, MD, Principal Investigator — Pauls Stradins Clinical University Hospital
Locations (1):
- Pauls Stradins Clinical University Hospital, Riga, Latvia

IPD SHARING:
Plan to Share IPD: No